CLINICAL TRIAL: NCT06762197
Title: Radial Extracorporeal Shockwave Versus Low Level Laser Therapy in Management of Patients With Chronic Piriformis Muscle Syndrome
Brief Title: Radial Shockwave Versus Low Level Laser Therapy in Patients With Chronic Piriformis Muscle Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mahdi Ali Ibrahim, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mohamed-004968
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Extracorporeal Shock Wave; Radial Shock Wave; Low Level Laser; Piriformis Muscle Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Extracorporeal Shockwave Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional program (Active Comparator): twenty one patients of chronic piriformis muscle syndrome will be treated by the conventional physical therapy program in the form of (hot packs, local massage and stretching exercise) for 6 weeks (two times per week).
  Interventions: Other: Conventional treatment
- Radial Extracorporeal shock wave (Experimental): twenty one patients of chronic piriformis muscle syndrome will be treated with Radial Extracorporeal shock wave in addition to the conventional physical therapy program in the form of (hot packs, local massage and stretching exercise) for 6 weeks (two times per week).
  Interventions: Other: Conventional treatment; Device: shockwave therapy
- low level laser therapy (Experimental): twenty one patients of chronic piriformis muscle syndrome will be treated with low level laser therapy in addition to the conventional physical therapy program in the form of (hot packs, local massage and stretching exercise) for 6 weeks (two times per week).
  Interventions: Other: Conventional treatment; Device: low level laser therapy

INTERVENTIONS:
Other: Conventional treatment — Physical therapy can be beneficial for patients with piriformis syndrome, including stretching exercises, local massage, and superficial heat. Traditional stretching techniques include external rotation, hip flexion, and adduction. A hot pack on the trigger point area for 10 minutes followed by passive stretching for 30 seconds each.
Device: shockwave therapy — Shockwave therapy is a non-invasive alternative treatment for muscle disorders like sports and traumatic injuries, as it reduces pain and promotes soft tissue repair. In a study, patients in group A were treated with three sessions of Storz Medical Shock Wave MP100, each consisting of 2000 pulses with a total energy dose of 1080 mJ / mm. The study aimed to determine the location of the piriformis muscle in the prone position.
  Arms: Radial Extracorporeal shock wave
Device: low level laser therapy — Low Level Laser Therapy, also known as Photo-biomodulation, is a low-intensity light therapy that triggers biochemical changes within cells, similar to photosynthesis in plants. It can treat nociceptive and neuropathic pain, but central pain has not been proven responsive to low level laser therapy.
  Arms: low level laser therapy

SUMMARY:
The study aims to compare the effects of radiation shockwave and low-level laser therapy on piriformis muscle thickness, lower extremity function, pain intensity, and hip range of motion in patients with piriformis syndrome.

DETAILED DESCRIPTION:
Low back pain affects 75%-84% of the general population in developed countries, with piriformis syndrome being more common in women. piriformis syndrome is a neuromuscular disorder caused by the compression of the sciatic nerve in the infra-piriformis canal, causing sciatic pain, tingling, and numbness. Few studies have examined the effectiveness of shockwave therapy in treating piriformis syndrome, but this study aims to compare results to improve treatment outcomes, save time and money, and add value to physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients' males and females with piriformis syndrome

  * Their age will range from 30-50 years old
  * Body mass index will be 25 to 30 (kg/m²).
* Both males and females.
* Low back pain radiating to posterior thigh, calf and Foot.
* Chronic piriformis syndrome due to micro trauma.
* Gluteal pain with or without radiation through sciatic nerve pathway.
* Faber test and Fair test and Beatty test positive.
* Diagnosed sub-acute and chronic piriformis syndrome.
* One-sided piriformis syndrome.
* Tenderness over lower back, buttocks and hip joint.

Exclusion Criteria:

- Piriformis syndrome due to macro trauma.

* Lumbo-sacral disc lesion and spinal stenosis.
* Lumbar spondylolisthesis.
* Pregnancy
* Recent fracture and surgery of spine, hip, knee and Ankle.
* Baker's cyst.
* Degenerative disease of spine and hip.
* Intermittent vascular claudication.
* Past history of vertebral fracture and spinal surgery
* Spinal tuberculosis.
* Rheumatoid disease.
* Disc pathology and mechanical back pain.
* Presence of malignant disease.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the change of body mass index | at baseline and after 6 weeks
  Weight and height Scale will be used to measure body mass index
assessing the change of pain intensity | at baseline and after 6 weeks
  The 10-cm visual analogue scale has been proven reliable, valid, and responsive for assessing pain levels, with 0 indicating no pain and 10 indicating the worst pain possible, demonstrating its effectiveness in measuring pain.

SECONDARY OUTCOMES:
assessing the change of functional status | at baseline and after 6 weeks
  The patient's functional status is assessed using the Lower Extremity Functional Scale before treatment. This self-assessment tool is valid and reliable, and the patient's score on the questionnaire is evaluated. The scale is free for clinical or research purposes.
assessing the change of range of motion of lower limb | at baseline and after 6 weeks
  Goniometer measurement is used to assess the range of motion of hip internal and external rotation before and after intervention. This simple test is accurate and reliable in detecting changes in hip range of motion, making it a valid measure to detect underlying hip pathology and enable surgical intervention based on it.
assessing the change of piriformis muscle thickness | at baseline and after 6 weeks
  Ultrasound guided measurement for piriformis M.sc thickness may be a reliable technique for early diagnosis of post-operative pain syndrome, increasing conservative treatment options and routinely evaluating patients with unidentified causes of buttock pain. The technique involves placing a probe in the patient's prone position, moving the patient's lower leg to confirm the piriformis position, and measuring piriformis thickness in the medial part of the ischium.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic in physiotherapy department at EL KATEB Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No